CLINICAL TRIAL: NCT03754205
Title: The Clinical, Histopathological, Cytological and Microbiological Efficacy of the Micro-ablative Fractional CO2 Laser : A Double-blind Randomized Placebo-controlled Trial
Brief Title: Vaginal CO2 Laser and the Genitourinary Syndrome of Menopause
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Themos Grigoriadis, Assistant Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 674/03-09-2018
Record Dates: First submitted 2018-10-28; First posted 2018-11-27 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Vaginal Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Group (Experimental): Microablative Fractional CO2 laser therapy at monthly intervals.
  The laser parameters that will be used are the following: (1) Power: 30 ή 40 watts, 2) Dwell time:1000μs, 3) Spacing 1000 μm, 4) Depth: SmartStak parameter from 1-3 depending on the treatment status, 5) D-pulse mode.
  Interventions: Device: Microablative Fractional CO2 laser
- Placebo Group (Placebo Comparator): Placebo CO2 laser therapies at monthly intervals.
  The laser parameters that will be used are the following: 1) Power: 0.5 watts, 2) Dwell time:1000μs, 3) Spacing 1000 μm, 4) Depth: SmartStak parameter 1, 5) Smart-pulse mode.
  Interventions: Device: Microablative Fractional CO2 laser

INTERVENTIONS:
Device: Microablative Fractional CO2 laser — 3 therapies intravaginally administered will be applied at monthly intervals
  Other Names: SmartXide2 V2LR, Monalisa Touch, DEKA, Florence, Italy

SUMMARY:
This study evaluates the clinical, histopathological, cytological and microbiological efficacy of Microablative Fractional CO2 laser intravaginally administered in postmenopausal women with Genitourinary Syndrome of Menopause. Half participants will receive active CO2 laser therapy, while the other half will receive placebo CO2 laser therapy.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of vaginal atrophy (dyspareunia and/or vaginal dryness)
* Menopause

Exclusion Criteria:

* Systemic or local hormonal therapy the last 6 months
* Use of moisturizers or lubricants the last month
* Active genital infection (i.e herpes, vaginitis)
* Prolapse stage >=2
* Underlying pathologies that could interfere with the protocol compliance

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-04-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
10-centimeter Visual Analogue Scale assessing intensity of dyspareunia and dryness | 24-months
  It is a straight line with 2 endpoints "0" and "10". Zero defines "no dyspareunia at all" and "no dryness at all" , while 10 "dyspareunia as bad as it could be" and "dryness as bad as it could be". Participants will draw a line at or between the 2 end points. The distance between zero and drawn line will define the intensity of dyspareunia and dryness

SECONDARY OUTCOMES:
Day-to Day Impact of vaginal aging questionnaire (DIVA) | 24 months
  It includes 4 domains: activities of daily living (5 items), sexual functioning (5 items), emotional well-being (4 items), self-concept and body image (5-items). Each item of each domain could receive values from 0 to 4. Mean scores are calculated on each of the domain scales. Higher scores indicate greater symptom impact
Patients Global Impression of Improvement | 24 months
  It is a single question with 7 possible answers. Patients will chose the answer that applies at their impression of improvement after the laser therapy
10-centimeter Visual Analogue Scale assessing intensity of itching, burning and dysuria | 24 months
  It is a straight line with 2 endpoints "0" and "10". Zero defines "no symptom at all", while 10 "symptom as bad as it could be" and "dryness as bad as it could be". Participants will draw a line at or between the 2 end points. The distance between zero and drawn line will define the intensity of symptom
3 days voiding diary | 24 months
  Assesses bladder function (frequency, urgency and incontinence)
Female Sexual Function Index | 24 months
  It includes 6 domains assessing sexual functioning (desire, arousal, orgasm, lubrication, satisfaction and pain). Total score is calculated by summing scores of the 5 domains multiplied by certain factors with a minimum value of 2 and maximum 36
International Consultation on Incontinence Questionnaire Short Form/Female Lower Urinary tract Symptoms (ICIQ-FLUTS) | 24 months
  It is a 12-items questionnaire evaluating nocturia, urgency, bladder pain, frequency, hesitancy, straining, intermittency, urinary incontinence (urge, stress and unexplained), frequency of urinary incontinence and nocturnal enuresis. Filling, voiding and incontinence symptoms subscales range from 0 to 15, 0 to 12 and 0 to 20, respectively.
King's Health Questionnaire (KHQ) | 24 months
  It has 3 sections: 1) general health and overall health related to urinary symptoms with 2 questions, 2) incontinence impact, role limitations, physical limitations, social limitations, personal limitations, emotions, sleep and energy, and severity coping measures with 19 questions and 3) bother or impact of urinary symptoms with 11 questions. Scores of each domain of the 2 sections range from 0 to 100. Scores of the third section range from 0 to 3. Higher scores indicate higher impact of urinary incontinence.
Vaginal Maturation Value | 24 months
  It is calculated by defining the percentage of superficial, intermediate and parabasal epithelial cells on the vaginal pap smear, following the formula (1x%superficial)+(0.5x%intermediate)+(0x%parabasal). It may receive values from 0 to 100%.It is considered to be an indicator of the estrogenic stimulation, whereas values of 0-49%, 50-64% and 65-100% indicate absent/low, moderate and high estrogenic effect on the vaginal epithelium, respectively.
Vaginal Health Index Score | 24 months
  It evaluates vaginal elasticity, fluid volume, ph of vaginal fluid, epithelial integrity and moisture. Each one of these may receive scores from 1 to 5. Total score is calculated by summing the 5 scores ranging from 5 to 25. Higher scores indicate better vaginal status.
Epithelial thickness | 24 months
  Biopsies will be obtained from the lateral vaginal wall. Epithelial thickness (in μ) will be measured by a vertical line between basal layer cells and superficial layers.
Number of Blood vessels | 24 months
  Computerized determination of number of capillary profiles in the test area will be performed percent of total area of subepithelial stroma), will be performed.
Size of blood vessels | 24 months
  Computerized determination of diameter (in μ), length (in μ) αnd width (in μ) will be performed.
Density of blood vessels | 24 months
  Computerized determination of volume density of blood vessels in percent of total area of subepithelial stroma will be performed
Cultures of vaginal samples | 24 months
  Lactobacilli, aerobic bacteria, anaerobic bacteria, fungi will be evaluated
Polymerase Chain Reaction | 24 months
  Lactobacilli, bacteria and fungi will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Athanasiou, Associate Proffesor, Principal Investigator — National and Kapodistrian University of Athens, Greece
Locations (1):
- Urogynecological Unit of Alexandra Hospital, Athens, Greece

REFERENCES:
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601